CLINICAL TRIAL: NCT05099770
Title: A Phase 3 Randomized Controlled Study of Renal Autologous Cell Therapy (REACT) in Subjects With Type 2 Diabetes and Chronic Kidney Disease (REGEN-006)
Brief Title: Proact: A Study of REACT in Subjects With Type 2 Diabetes Mellitus and Chronic Kidney Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Prokidney (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REGEN-006
Record Dates: First submitted 2021-10-18; First posted 2021-10-29 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes Mellitus; Chronic Kidney Diseases
Keywords: REACT®; Type 2 Diabetes Mellitus; Rilparencel; Proact
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sham Procedure (Sham Comparator): Participants randomized to the Sham Comparator arm will have 2 sham procedures.
  Interventions: Procedure: Sham Comparator
- Experimental (REACT/rilparencel injections) (Experimental): Participants randomized to the experimental arm will receive 2 injections of REACT/ rilparencel.
  Interventions: Biological: Renal Autologous Cell Therapy (REACT)

INTERVENTIONS:
Biological: Renal Autologous Cell Therapy (REACT) — Participants will have a kidney biopsy followed 14 weeks later with a REACT injection into the biopsied kidney, then, another 12 weeks (+28 days) later a REACT injection into their contralateral kidney.
  Arms: Experimental (REACT/rilparencel injections)
Procedure: Sham Comparator — Participants will have 2 sham procedures that simulate real biopsy and injection procedure. No tissue is taken during biopsy and nothing is injected into kidney. The second sham procedure will occur 12 weeks (+28 days) after the first sham procedure.
  Arms: Sham Procedure

SUMMARY:
The purpose of this study is to assess the safety and efficacy (including durability) of up to 2 REACT/rilparencel injections given 12 weeks (-14 days to +28 days) apart and delivered percutaneously into biopsied and non-biopsied contralateral kidneys in participants with T2DM and CKD.

DETAILED DESCRIPTION:
Randomized multi-center, blinded intervention, two cohort, study whereby eligible participants will be randomized 1:1, prior to kidney biopsy, to 1 of 2 cohorts. Cohort 1 participants will have scripted sham procedures that mimic the sounds and activities of biopsy, injection procedures, and evaluations as a control for Cohort 2 participants who will have a kidney biopsy followed 12 weeks later with a rilparencel injection into the biopsied kidney, then, another 12 weeks later, a rilparencel injection into the contralateral kidney. All participants will be followed to the global trial end date. This event driven study is estimated to have a total maximum duration of 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is male or female, 30 to 80 years of age on the date of informed consent.
2. Documented diagnosis of type 2 diabetes mellitus (T2DM) and chronic kidney disease as the underlying cause of kidney disease (diagnosis does not have to be confirmed by kidney biopsy).

   1. eGFR of at least 20 mL/min/1.73 m2 AND <30 mL/min/1.73 m2, not requiring kidney dialysis. UACR level cannot exceed 5000 mg/g (565 mg/mmol), OR
   2. eGFR of 30 to ≤ 35 mL/min/1.73m2 AND UACR of 300 to ≤ 5000 mg/g (33.9 mg/mmol to ≤565 mg/mmol).
3. Serum glycosylated hemoglobin (HbA1c) of 9.5% or lower at Screening.
4. Systolic blood pressure of ≤ 140 mm Hg and diastolic blood pressure of ≤ 90 mm Hg at Screening, based on average of 3 consecutive measurements obtained seated or supine. Note: Retesting may be performed if initial screening blood pressure exceeds eligibility criteria for systolic and/or diastolic blood pressure. Changes in blood pressure Page 46 of 113 CONFIDENTIAL ProKidney Renal Autologous Cell Therapy Clinical Protocol REGEN-006 USAN/INN: Rilparencel Version 6.0 medications will be recorded in the appropriate eCRF. (refer to BP procedures)
5. All participants should be strongly considered for treatment with sodium-glucose cotransporter 2 inhibitor (SGLT2i). For participants on SGLT2i medications, the dose must be stable for at least 4 weeks prior to randomization. Note: The reason for a participant NOT receiving SGLT2i therapy at the time of randomization will be documented in the eCRF. (See Section 7.1 for additional guidance about Concomitant Therapies).
6. On a clinically relevant, maximally tolerated dose of an angiotensin converting-enzyme inhibitor (ACEI) OR an angiotensin receptor blocker (ARB), unless not tolerated or contraindicated. The dose must be stable for at least 4 weeks prior to randomization. Note: The reason for a participant NOT receiving an ACEI or ARB at the time of randomization will be documented in the eCRF. (See Section 7.1 for additional guidance about Concomitant Therapies).
7. Participant agrees, and in the judgement of the Investigator, is able to refrain from using therapies that may increase bleeding risk for the specified pre-procedure and postprocedure (biopsy/sham biopsy and rilparencel/sham injections) durations in the discretion of the PI in consultation with the treating physician, in accordance with the required minimum medication-specific guidelines for high-risk procedures59 and patients with advanced CKD.

   * Nonsteroidal anti-inflammatory drugs (NSAIDS) such as ibuprofen and naproxen
   * Aspirin
   * Platelet aggregation inhibitors (PAIs) such as clopidogrel, prasugrel, and dipyridamole
   * Factor Xa inhibitors
   * Warfarin
   * Heparin products
   * Other anticoagulation.
8. Participant is willing and able to cooperate with all aspects of the protocol.
9. Participant is willing and able to provide signed informed consent.

Exclusion Criteria:

1. The participant has a history of type 1 diabetes mellitus.
2. The participant has a history of renal transplantation or other organ transplantation (corneal transplants are not an exclusion), solitary kidney, recurrent complicated urinary tract infections or complicated kidney stones. Urinary tract infections identified prior to renal biopsy or injection should be resolved prior to procedures.
3. The participant has any other known underlying cause of kidney disease, including but not limited to: Autosomal dominant and recessive polycystic kidney disease, primary focal segmental glomerulosclerosis, vasculitis related CKD, IgA nephropathy and other immune modulated nephropathies, drug-induced CKD or other types of CKD or anatomic variants as determined by the Investigator or Sponsor that would interfere with biopsy and rilparencel injection procedure or confound study assessments.

   Note: The following are not considered exclusionary under the following conditions: (Unique situations should be discussed with the study Medical Monitor.)
   * Concomitant hypertension-related CKD
   * Anatomic abnormalities and benign conditions are not exclusionary if the kidney has accessible kidney cortex for biopsy and injection procedures and meets the criteria to receive the rilparencel injection.
   * Abnormalities on kidney biopsy (e.g., secondary focal segmental glomerulosclerosis) which are considered secondary to diabetes with the following conditions: lack of other identifiable etiology, full evaluation for other etiologies, no specific treatment administered other than diabetes management.
4. History of acute kidney injury or major surgery (based on the judgement of the Investigator and Medical Monitor) within 3 months prior to the Screening Visit.
5. Myocardial infarction, unstable angina, revascularization procedure (e.g. stent or bypass graft surgery), or cerebrovascular accident within 12 weeks before randomization, or a revascularization procedure is planned during the trial.
6. Current or history of heart failure of New York Heart Association (NYHA) Class IV cardiac disease.
7. History of malignancy within the past 3 years prior to Screening, except for basal cell and/or squamous cell carcinomas of the skin with apparent successful curative therapy, carcinoma of the cervix in situ, or a malignancy that in the opinion of the Investigator, along with agreement from the Medical Monitor, is considered treated with no evidence of disease and at minimal risk of recurrence.
8. Documented clinically significant liver disease, including acute or chronic hepatitis B or hepatitis C. Note: At the discretion of the Investigator, a participant who gives a history of a treated and cured Hepatitis C infection may be screened with a test for viral ribonucleic acid (RNA), and if a cure is demonstrated, the participant may be enrolled.
9. Known infection with HIV, active syphilis, or other unresolved active genitourinary infection, or active tuberculosis requiring treatment at Screening.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 685 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Clinical Endpoint | up to 60 Months
  The time from first injection to the earliest of:
  * At least 40% reduction in eGFR, sustained for 30 days, OR
  * eGFR <15 mL/min/1.73m², sustained for 30 days and/or chronic dialysis, and/or kidney transplant OR
  * Renal or cardiovascular death

SECONDARY OUTCOMES:
Secondary Composite Endpoint: Change in eGFR from first injection | up to 60 Months
  • Time from first injection to at least a 40% reduction in eGFR sustained for 30 days.
Secondary Composite Endpoint: Change in eGFR from first injection to End Stage Renal Disease (ESRD) | up to 60 Months
  • Time from first injection to eGFR < 15 mL/min/1.73m² sustained for 30 days and/or chronic dialysis, and/or kidney transplant.
Secondary Composite Endpoint: Mortality | up to 60 Months
  The time from first injection to all-cause mortality.
Secondary Composite Endpoint: Quality of Life Changes | up to 60 Months
  • Changes from Baseline in patient-reported outcome from the Burden of Kidney Disease domain at Week 52 from the Kidney Disease Quality of Life (KDQOL) Questionnaire.
  The survey is used to assess the burden, symptoms/problems, and effects of kidney disease on a patient's quality of life.
Secondary Composite Endpoint: Quality of Life | up to 60 Months
  Changes from Baseline in patient-reported outcome EuroQol 5-Dimension 5-Level (EQ5D-5L) at Week 52.
  The descriptive system is divided into 5 levels of perceived problems with level 1 (indicating no problem) and level 5 (indicating extreme problems).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Prokidney
Locations (86):
- United States (71):
  - University of Arizona, Tucson, Arizona
  - Amicis Research Center, Beverly Hills, California
  - Paradise Clinical Research Group LLC, Glendora, California
  - Kidney Consultants Medical Group, Granada Hills, California
  - IMD Clinical Trials, Huntington Park, California
  - Advanced Medical Research, LLC, Lakewood, California
  - Medicine and Nephrology Associates, Los Alamitos, California
  - Academic Medical Research Institute, Los Angeles, California
  - Southern California Hospital, Los Angeles, California
  - Allameh Medical Corporation, Mission Viejo, California
  - Golden Pacific Nephrology Medical Clinic Inc, Monterey Park, California
  - Northridge Kidney Care Center, Northridge, California
  - Valley Renal Medical Group, Northridge, California
  - Valley Clinical Trials, Northridge, California
  - Integrity Medical Discovery, Pico Rivera, California
  - Nephrology Associates Medical Group, Riverside, California
  - UC Davis Medical Group GI Unit, Sacramento, California
  - North America Research Institute, San Dimas, California
  - Henry Mayo Newhall Hospital, Valencia, California
  - Nephrology Associates PA, Newark, Delaware
  - West Broward Research Institute, Coral Springs, Florida
  - Florida Kidney Physicians, Fort Lauderdale, Florida
  - South Fort Lauderdale Nephrology, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Ethos Palm Beach, Loxahatchee Groves, Florida
  - Global Clinix, LLC, Miami, Florida
  - Professional Research Center, Inc., Miami, Florida
  - New Phase Clinical Trials, Miami Beach, Florida
  - Infigo Clinical Research, Sanford, Florida
  - Genesis Clinical Research, Tampa, Florida
  - American Clinical Trials, Acworth, Georgia
  - Boise Kidney and Hypertension PLLC, Boise, Idaho
  - Care Institute, Chubbuck, Idaho
  - Insight Hospital & Medical Center Chicago, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - Indiana Nephrology, Fishers, Indiana
  - University of Iowa, Iowa City, Iowa
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Washington Nephrology Associates, Takoma Park, Maryland
  - Holyoke Medical Center, Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Nephrology Center, PC, Kalamazoo, Michigan
  - St. Clair Nephrology Research, Roseville, Michigan
  - Nephrology and Hypertension Associates, Tupelo, Mississippi
  - Saint Louis University, St Louis, Missouri
  - Nevada Kidney Disease & Hypertension Center, Las Vegas, Nevada
  - Seacoast Kidney & Hypertension Specialists, Portsmouth, New Hampshire
  - ICAHN School of Medicine at Mount Sinai, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Lifespan Clinical Research Center, East Providence, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Dunes Clinical Research, Dakota Dunes, South Dakota
  - Knoxville Kidney Center, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Pioneer Research Solutions, Inc., Cypress, Texas
  - Texas Tech Health Sciences, El Paso, Texas
  - Texas Tech University Health, El Paso, Texas
  - Plaza Nephrology, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Prolato Clinical Research Center, Houston, Texas
  - Clinical Research Strategies, Inc, Houston, Texas
  - United Memorial Medical Center, Houston, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - University Health System, San Antonio, Texas
  - Prolato Clinical Research Center - Sugar Land, Sugar Land, Texas
  - Renal Physicians of Montgomery County, The Woodlands, Texas
  - Salem VA Medical Center, Salem, Virginia
  - Providence Medical Research Ctr, Spokane, Washington
  - University of Wisconsin-Madison, Madison, Wisconsin
- St. George Hospital, Kogarah, New South Wales, Australia
- Lakeridge Health Corporation-Oshawa, Oshawa, Ontario, Canada
- Mexico (2):
  - "Ignacio Chavez" National Cardiology Institute, Tlalpan, Mexico City
  - National Institute of Medical Sciences and Nutrition Salvador Zubiran, Tlalpan, Mexico City
- Puerto Rico (2):
  - Torre Medica San Lucas, Ponce
  - San Miguel Medical, Trujillo Alto
- Taiwan (8):
  - Far Eastern Memorial Hospital, New Taipei City
  - Taipei Medical University - Shuang Ho Hospital, Ministry of Health and Welfare, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Taipei Medical University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taipei Municipal Wanfang Hospital Managed by Taipei Medical University, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei
- Royal London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cizman B, Butler EL, Stavas J, Prakash R, Saad T, Silva A, Wooldridge T, Aqeel A, Yan H, Barysauskas CM, Culleton B. A Randomized Clinical Trial of Kidney Autologous Cell Therapy in Diabetic Kidney Disease. Clin J Am Soc Nephrol. 2026 Jan 2. doi: 10.2215/CJN.0000000969. Online ahead of print. No abstract available. PMID 41481370
- [Derived] Patel HA, Wang J, Zinn CJ, Learmonth M, Lerman LO, Wolfram J, Hickson LJ. Fortifying the Diabetic Kidney Disease Treatment Armamentarium: Multitarget Senotherapeutic and Regenerative Strategies. J Am Soc Nephrol. 2025 May 7;36(8):1655-1658. doi: 10.1681/ASN.0000000754. No abstract available. PMID 40333016